CLINICAL TRIAL: NCT00585182
Title: Venous Thromboembolism Prevention in the Morbidly Obese Medically Ill Patient: A Pharmacological Analysis of the Predictability of Prophylactic Weight-Based Enoxaparin Dosing.
Brief Title: Study to Evaluate Weight-based Enoxaparin Dosing in Obese Medical Patients at Risk for DVT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20115; Utah IRB 20115
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Venous Thrombosis; Anticoagulants
Keywords: Obesity; venous thrombosis; Anticoagulants
MeSH Terms: conditions — Obesity; Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Enoxaparin 0.5 mg/kg once daily

INTERVENTIONS:
Drug: Enoxaparin 0.5 mg/kg once daily — Enoxaparin 0.5 mg/kg (kg= actual body weight) subcutaneous once daily for 2 doses.
  Other Names: Lovenox

SUMMARY:
Deep vein thrombosis(DVT) is a common complication in hospitalized medical patients. Consensus guidelines recommend using medications such as heparin or low-molecular-weight heparins (LMWH) to prevent DVT in these patients. Generally, these medications are given in a fixed dose that is the same for everyone. The appropriate dose of medication in patients with severe obesity is uncertain. There is some evidence that the use of standard fixed-doses in severely obese patients may not provide adequate protection against DVT. The purpose of this study is to evaluate a weight-based dose(0.5 milligrams per kilogram of body weight) of the commonly prescribed LMWH, enoxaparin in severely obese patients to determine if predictable levels of blood thinning can be achieved. We hypothesize that dosing enoxaparin 0.5mg/kg once daily in severely obese patients will lead to predictable blood levels.

DETAILED DESCRIPTION:
Background and Introduction:

Venous thromboembolism (VTE) is a significant cause of morbidity and mortality in hospitalized patients. It is a well-known complication in patients after major surgery or trauma. More recently, medically ill patients have been identified as another high risk group with up to 15% of patients experiencing VTE in the absence of prophylaxis. 1 Several studies have found the use of enoxaparin, dalteparin, and fondaparinux to be safe and effective in reducing risk of VTE by 45% to 63% in medically ill patients. 1-3 Additionally, enoxaparin has been found to be at least as safe and effective as unfractionated heparin for VTE prophylaxis. 4 Enoxaparin 40 mg once daily has been shown to be a safe and effective prophylactic therapy in hospitalized patients. 1

In thromboprophylaxis studies, including those investigating enoxaparin 40 mg once daily, morbidly obese patients (greater than or equal to 35 kg/m2) have been grossly under-enrolled. This is problematic for several reasons. First, the drug distribution is weight dependent and therefore, anticoagulant levels will differ according to a patient's weight. 5 Secondly, the FDA approved doses are fixed doses that do not take into account body weight. Thirdly, obese patients are at greater risk for failure in preventing VTE and obese patients are probably at greater risk for developing VTE. 6 Lastly, morbidly obese patients are becoming quite common as the population as a whole is becoming more obese.

Even with this information, there are no standards of VTE prophylaxis in obese patients. Optimal means of delivering safe and effective thromboprophylaxis in this group is unknown. When using LMWH's, consensus recommendations have been to monitor peak anti-Xa activity targeting a level of 0.1-0.2 units/mL. 5 However, many hospitals do not have access to anti-Xa monitoring. Studies evaluating the predictability of weight-based prophylactic dosing of tinzaparin have demonstrated that anti-Xa levels are predictably achieved and therefore, laboratory monitoring may not be necessary with this dosing strategy.7 However, tinzaparin is not widely utilized in the U.S. and uncertainties remain about whether predictable anti-Xa levels can be achieved with a weight-based prophylactic regimen using the more commonly used drug enoxaparin. If weight-based dosing with enoxaparin is shown to result in predictable anti-Xa activity in obese patients, the need for monitoring would be obviated.

Objectives: The primary objective is to evaluate the predictability in achieving target anti-Xa activity levels in morbidly obese medically ill patients using weight-adjusted (0.5 mg/kg) once daily prophylactic dose of enoxaparin. The secondary objective is to gain information to evaluate the pharmacokinetic curve of enoxaparin in obese patients over 18 hours after the second dose.

Participant Selection Criteria: VTE risk will be evaluated with an institutionally utilized risk stratification scheme. This risk stratification scheme which was drafted by a multi-disciplinary panel, represents standard of care for medically ill patients at the University of Utah.

Inclusion Criteria: Medically ill patients who are greater than 18 years of age who have a body mass index (BMI) greater than or equal to 35 kg/m2 who are admitted to the University of Utah Medical Center, are at risk for VTE, and are eligible for pharmacological prophylaxis as determined by patient's provider will be consented for the study.

Exclusion Criteria: Patients who are pregnant (a urine HCG will be performed if a female of child-bearing age is not on reliable birth control, or if otherwise clinically indicated), are currently on therapeutic anticoagulation, have a bleeding disorder, platelet count of less than 100,000/mL, coagulopathy, active bleeding, creatinine clearance less than 30 mL/min (based on Cockcroft-Gault equation, and rounding serum creatinine to 1 in patients greater than 65 years), or recent (within 14 days) stroke, surgery or trauma will be excluded.

Design: This is a single arm study enrolling consecutive eligible patients admitted to the University of Utah Medical Center. This is a descriptive study evaluating the feasibility and predictability of administering weight-adjusted enoxaparin (0.5mg/kg once daily) to achieve recommended target peak anti-Xa levels in patients at extreme body weight. The hypothesis is that weight-adjusted prophylaxis will reliably achieve recommended target anti-Xa levels. If so, this would obviate the future need for routine anti-Xa monitoring using this pharmacologic regimen.

Additionally, there will also be a parallel cohort evaluating a day 2 pharmacokinetic curve by 5-serial anti-Xa activity measurements in a subset of up to 2-3 patients in each weight group.

Study procedures: Consecutive eligible patients will be enrolled if informed consent is given. Consent will be obtained in the University Hospital, mainly on the Internal Medicine Floor. It will be obtained by the one of the study co-investigators. At least one person who is obtaining consent will be available to consent patients any time of day and will have adequate time to exchange information and answer questions between investigator and participant.

The study protocol uses a VTE prevention regimen that employs rational pharmacologic principles and is in line with published recommendations for prophylaxis in this patient population. In consideration of having a comparator cohort group, we would consider it to be unethical to have a cohort group receiving enoxaparin 40 mg subcutaneously once daily as a comparator group because pharmacologic data strongly suggests that effective levels of anticoagulation would not be achieved in this population of patients. 8 Informed consent was felt optimal in order to allow patients to fully understand that this regimen, although it is an acceptable standard of care, is being employed under the broader context of a study whereby other patient data will be collected and recorded in prospective fashion. Once informed consent is obtained, patients will begin VTE prophylaxis with enoxaparin 0.5 mg/kg subcutaneously once a day. Peak anti-Xa activity will be obtained in all patients through a venipuncture 4-6 hours after the first or second dose has been given. Five milliliters of blood will be drawn. This is the amount of blood that is needed for this laboratory test to be performed. Baseline clinical and demographic information will be obtained and recorded on standard case reporting forms, CRF (see Appendix B). Patients will continue prophylaxis as deemed necessary by their attending physician through the duration of their hospital stay or unless dictated otherwise by the patient's attending physician. Adverse events such as VTE, bleeding event, or thrombocytopenia will be recorded during the hospital stay (see Appendix C).

If patients consent to do the additional testing, this will be marked on the consent form. These patients will have anti-Xa levels drawn before the first enoxaparin dose, and then at 4h, 6h, 12h, and 18h after the second dose of enoxaparin. If the 12h anti-Xa level is obtained and is less than 0.05 units/mL, then the 18 hour blood test can be eliminated. The purpose of this section is to provide us with information to evaluate the pharmacokinetic curve of enoxaparin in obese patients over 18 hours.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (BMI>35kg/m2)>18 years of age admitted to medical service and considered at increased risk for DVT and whom pharmacological prophylaxis is being considered by treating physician.

Exclusion Criteria:

* Pregnancy
* Currently on alternate therapeutic anticoagulant (warfarin, heparin, LMWH)
* Platelet count <100,000, CrCl <30ml/min, or coagulopathy
* recent (within 14 d) stroke, trauma, or major surgical procedure
* Active bleeding or deemed at increased bleeding risk by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Pendleton, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 patients met eligibility criteria and completed the protocol enrolled from the University of Utah Hospital Inpatient Medical Service
Period: Overall Study
Arm/Group | Enoxaparin 0.5mg/kg Once Daily
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enoxaparin 0.5mg/kg Once Daily
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Peak Low Molecular Weight Heparin Anti-Xa Activity Level.
Description: The Rotachrom® assay using the STA-Compact instrument (Diagnostica Stago, Parsippany, NJ) was used to quantitate anti- Xa (LMWH) activity for enoxaparin. The sensitivity of this assay is 0.2 U/mL and within run imprecision is 5.5 (% CV) at 1 U/mL. The assay is linear between 0.2-2.0 U/mL
Time Frame: 4 - 6 hours after enoxaparin dosing on Day 1 and Day 2
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Enoxaparin 0.5mg/kg Once Daily
Number analyzed (Participants) | 28
IU/mL | 0.25 (0.11)

2. Secondary Outcome: Clinically Relevant Bleeding Events
Description: Clinically Relevant Bleeding is defined as fatal bleeding, symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells, or bleeding requiring intervention
Time Frame: Participants were followed for the duration of hospital stay, an average of 5 days
Measure: Number; unit: Events
Arm/Group | Enoxaparin 0.5mg/kg Once Daily
Number analyzed (Participants) | 28
Events | 0

ADVERSE EVENTS:
Arm/Group | Enoxaparin 0.5mg/kg Once Daily
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
This study was limited by a relatively small sample size, lack of long-term clinical outcome data, and the use of only a single anti-Xa level, rather than repeat measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No